CLINICAL TRIAL: NCT04312776
Title: Tracing MRSA in Households With Patients Infected With CA-MRSA by WGS
Status: Completed | Type: Observational
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-cang Zhou M.D., Prof., Sir Run Run Shaw Hospital
Other Study IDs: SRRSH-Household01
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: MRSA
Keywords: MRSA; Whole-genome sequencing

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients infected with CA-MRSA: It is an observational study, no interventions to any of the two study arms.
  Interventions: Other: none intervention
- Healthy people without any infection: It is an observational study, no interventions to any of the two study arms.
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention

SUMMARY:
From the 1980s to the late 1990s, highly toxic methicillin-resistant Staphylococcus aureus (MRSA) strains (called community-associated [CA] MRSA) appeared in the community. Although the prevalence of HA-MRSA (health-related MRSA) infection remained stable between 1998 and 2008, the CA-MRSA (community-related MRSA) infection rate increased. By far, the most common manifestations of CA-MRSA related diseases are skin and soft tissue infections. Skin and soft tissue infections (SSTIs) account for at least 90% of CA-MRSA infections. CA-MRSA strains also cause bone and joint infections, such as osteomyelitis and respiratory infections, such as pneumonia, sepsis, and urinary tract infections. Given that Staphylococcus aureus can live in the home as a settler or environmental pollutant, the environment can be used as a medium for obtaining and transmitting MRSA. In addition, transmission of MRSA between pets and humans has been proposed, but the directionality is unclear. In this study, we report an in-depth epidemiological and genomics study of a community-associated methicillin-resistant Staphylococcus aureus infection in SSRSH, Zhejiang Province, China.

DETAILED DESCRIPTION:
Eligibility criteria:

1. Inclusion criteria: Patients (Child, Adult) with infections caused by S. aureus from the sites as follows: blood stream, skin or soft tissue, cerebrospinal fluid, bone and joint, genitourinary tract, infection of indwelling intravascular device, surgical wound, respiratory tract (organism grown from sputum and infiltrate on chest X-ray), peritoneal fluid or other otherwise sterile body fluids.
2. Exclusion criteria: Patients with risk factors for nosocomial or medically related infections, and patients who have been decolonized (using mupirocin, chlorhexidine or bleach) in the past month.

Outcome measures:

1. Isolation rate of staphylococcus aureus and methicillin-resistant staphylococcus aureus on domestic environment, contact and pets and livestock.
2. Molecular characteristics of CA-MRSA isolates recovered in Chinese hospitals, home environments, contacts, and pets and livestock.

Definition:

A MRSA infection was considered to be HA-MRSA by the CDC epidemiologic definitions if, in the year prior to culture, the subject had surgery, hospitalization, hemodialysis or a stay in a long-term care facility, if an indwelling vascular catheter was in place at the time of culture, or if the subject was an inpatient hospitalized for 2 days at the time of culture. Otherwise, the subject was considered to have a CA-MRSA infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients (Adult) with infections caused by S. aureus from the sites as follows: blood stream, skin or soft tissue, cerebrospinal fluid, bone and joint, genitourinary tract, infection of indwelling intravascular device, surgical wound, respiratory tract (organism grown from sputum and infiltrate on chest X-ray), peritoneal fluid or other otherwise sterile body fluids.

Exclusion Criteria:

* Patients with risk factors for nosocomial or medically related infections, and patients who have been decolonized (using mupirocin, chlorhexidine or bleach) in the past month.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: No special requirements
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Clonal Distribution of CA-MRSA in China The distribution of sequence types in CA-MRSA isolates from China | During the study period (One years)

CONTACTS AND LOCATIONS:
Overall Officials: Yun-song Yu, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Sir Run Run Shaw Hospital, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided